CLINICAL TRIAL: NCT01932944
Title: Evaluation of the Accuracy of the Abbott Sensor Based Interstitial Glucose Monitoring System Compared to Venous and Capillary Glucose
Brief Title: Accuracy Characterization Study
Acronym: ACS
Status: Completed | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC13-126
Record Dates: First submitted 2013-08-28; First posted 2013-08-30 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Type2 Diabetes; Type1diabetes; Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment
  Interventions: Device: No treatment

INTERVENTIONS:
Device: No treatment

SUMMARY:
To demonstrate point accuracy of the Abbott Sensor Based Glucose Monitoring System (System) interstitial glucose results against venous glucose reference and capillary fingerstick using the Consensus Error Grid over the wear duration. During the course of the wear duration, the subject is required to be testing fingerstick glucose measurement at least 8 times a day for capillary reference glucose measurements and three in-clinic visits of maximum 10 hours each for venous reference glucose measurements. With every reference measurement, the subject or study staff will perform a measurement on the System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must have type 1 or type 2 diabetes for at least 2 years prior to enrollment.
3. Subject must require insulin therapy through an insulin pump and/or multiple daily insulin injections (at least 3 injections daily) for at least 6 months prior to enrollment.
4. Subject must be able to read and understand English.
5. In the Investigator's opinion, the Subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
6. Subject must be available to participate in all study visits up to a period of 14 days.
7. Subject must be willing and able to provide written signed and dated informed consent.

Exclusion Criteria:

1. Subject has known allergy to medical grade adhesive or isopropyl alcohol used to disinfect skin.
2. Subject is pregnant, attempting to conceive or not willing and able to practice birth control during the study duration.
3. Subject has skin lesions, scarring, redness, infection or edema at the application sites that could interfere with device placement or the accuracy of interstitial glucose measurements.
4. Subject currently is participating in another clinical trial.
5. Subject has donated blood within 112 days prior to the beginning of the study activities.
6. Subject has concomitant medical condition which, in the opinion of the Investigator, could interfere with the study or present a risk to the safety or welfare of the Subject or study staff. Such conditions include but are not limited to:

   * History of HIV, Hepatitis B or C, or other blood-borne pathogen;
   * Subject has an increased risk of bleeding.
   * Subject has X-ray, MRI or CT appointment scheduled during the period of study participation, and the appointment cannot be rescheduled for a time before study participation starts or after study participation ends.
   * Subject is unsuitable for participation due to any other cause as determined by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 1 or type 2 diabetes requiring multiple daily insulin injections (MDI) or continuous subcutaneous insulin infusion (CSII). No more than 10 subjects (5 per site) will have HbA1c > 8.5%, and no more than 10 subjects (5 per site) will have HbA1c < 7% based on the subject screening.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Accuracy of the Abbott Sensor Based Interstitial Glucose Monitoring System compared to venous and capillary glucose | 14 days
  To demonstrate point accuracy of the Abbott Sensor Based Glucose Monitoring (GM) System interstitial glucose results against venous glucose reference (YSI) using the Consensus Error Grid.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Christiansen, M.D., Principal Investigator — Diablo Clinical Research; Leslie Klaff, M.D., Principal Investigator — Rainier Clinical Research Center
Locations (2):
- United States (2):
  - Diablo Clinical Research, Walnut Creek, California
  - Rainier Clinical Research Center, Rainier, Washington